CLINICAL TRIAL: NCT00918944
Title: EHR Decision Support to Improve Outpatient Asthma Care
Brief Title: Electronic Health Record (EHR) Decision Support to Improve Outpatient Asthma Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2005-11-4596
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Asthma
Keywords: clinical decision support tool; electronic health record; control tool; spirometry; quality of life survey; provider survey
MeSH Terms: conditions — Asthma | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (Other): Practices with the EHR implemented will be randomized have the asthma disease management tools available passively (the control group).
  Interventions: Other: Control
- Intervention arm (Other): The intervention sites will have decision support alerts and reminders activated to guide providers toward these tools in the appropriate situations.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Control — The asthma disease management toolkit available to all practices in the EHR will consist of four elements:
  * A data entry tool for capturing asthma control data
  * Standardized documentation templates to facilitate severity classification
  * Order sets to facilitate ordering controller medications
  * An asthma care plan that can be supplied to families
  Arms: Control arm
Other: Intervention — Three alerts and two reminders will be programmed:
  * Alert providers to enter asthma severity classification if none is on file
  * Alert providers to prescribe controller medications for persistent asthma if none on file
  * Alert providers to complete an asthma care plan if none on file
  * Remind providers to review the asthma care plan if it is already on file by providing a link to the form
  * Remind providers that educational content is available on-line by providing a web link
  Arms: Intervention arm

SUMMARY:
To determine whether an innovative clinical decision support system embedded in an existing electronic health record (EHR) will improve provider adherence to the existing National Asthma Education and Prevention Program (NAEPP) guidelines.

12 primary care pediatric practices at The Children's Hospital of Philadelphia(both urban and suburban sites) will be randomized to receive either a passive EHR (control sites) or an interactive decision support system (intervention sites).

DETAILED DESCRIPTION:
After receiving a standardized education module based on NAEPP guidelines, 12 primary care pediatric practices (both urban and suburban sites) will be randomized to receive either a passive EHR (control sites) or an interactive decision support system (intervention sites).

The primary outcome of interest will be the proportion of patients on appropriate asthma controller medication compared over time. Secondary outcomes include the proportion of asthma patients with: 1) an updated asthma action plan 2) documentation of spirometry performed (6 to 17 yrs) and 3) an updated problem list reflecting current asthma severity. After hours calls to providers and types of office visits related to asthma will be tracked. 4) In addition, measurement of asthma-related quality of life and missed school and work in a sample of 200 subjects from each group will be performed. Contextual factors at the clinic and patient level will be examined to assess their association with outcomes of interest.

If shown to be successful, this type of clinical decision support, embedded within the EHR, has the potential to be a powerful tool to improve the implementation of asthma guidelines and clinical practice guidelines for other conditions and illnesses in the primary setting.

ELIGIBILITY:
Inclusion Criteria:

* Known patients with asthma

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-01; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the proportion of persistent asthmatic patients with at least one prescription for a controller medication in each period. There are two periods of study: baseline and intervention. | 6 months

SECONDARY OUTCOMES:
Secondary outcomes include the proportion of persistent asthmatic patients with 1)an updated asthma action plan, 2)spirometry as needed 3)problem list with current asthma severity 4)asthma-related quality of life scores 5)absent school and work days. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Louis M Bell, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States